CLINICAL TRIAL: NCT02542488
Title: Use of the STOPBANG Questionnaire for Predicting Obstructive Sleep Apnoea in Pregnancy
Brief Title: STOPBANG As A Screening Tool for Obstructive Sleep Apnoea in Pregnancy
Status: Completed | Type: Observational
Sponsor: City Hospitals Sunderland NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STOPBANGPREG
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Obstructive Sleep Apnoea; Pregnancy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women with BMI >39 at booking: All women will receive routine care and in addition will complete the 8 question STOPBANG screening tool, an Epworth sleepiness scale and have overnight oximetry recorded.
  Interventions: Other: STOPBANG Questionnaire; Diagnostic Test: Overnight pulse oximetry; Other: Epworth Sleepiness Scale

INTERVENTIONS:
Other: STOPBANG Questionnaire — 8 question screening tool comprised of the following questions:
  S: Do you Snore loudly? T: Do you often feel tired during daytime? O: Has anyone observed you stop breathing during your sleep? P: Do you have high blood pressure? B: Is your BMI >35 kg/m2? A: Are you >50 years old? N: Is your neck circumference >40cm? G: Is your gender male?
Diagnostic Test: Overnight pulse oximetry — All participants will be given a Masimo Rad8 pulse oximeter to take home and apply to their finger overnight to measure their heart rate and oxygen saturations while they sleep.
Other: Epworth Sleepiness Scale — A questionnaire that rates how tired they are doing everyday tasks

SUMMARY:
This study evaluates the use of the STOPBANG questionnaire to predict whether a pregnant woman with class III obesity has obstructive sleep apnoea. All participants will have a STOPBANG score and modified STOPBANG score (substituting Epworth score > 10 with the tired item) calculated and then be tested with overnight pulse oximetry to see if they meet ODI criteria for obstructive sleep apnoea.

DETAILED DESCRIPTION:
Obstructive sleep apnoea (OSA) is a condition in which the muscles and soft tissues of the throat collapse during sleep, resulting in them stopping breathing for a short period. It affects around 4% of all pregnant women and is more common in obese people. Pregnant women with untreated OSA are more likely to have pregnancy complications and are more likely to need a caesarean section. Babies born to mothers with untreated OSA are more likely to need neonatal treatment. If OSA is diagnosed and treated then these risks are reduced. In non-pregnant patients presenting for surgery, an screening tool called STOPBANG has been proven to be effective in identifying patients with OSA.

S: Do you Snore loudly? T: Do you often feel tired during daytime? O: Has anyone observed you stop breathing during your sleep? P: Do you have high blood pressure? B: Is your BMI >35 kg/m2? A: Are you >50 years old? N: Is your neck circumference >40cm? G: Is your gender male?

The investigators aim to assess whether STOPBANG can be used to identify OSA in obese pregnant women.

The aim is to recruit 100 pregnant women with a body mass index (BMI) ≥40 at Sunderland Royal Hospital. Data will be collected when they attend for their anomaly scan or glucose tolerance test (during the second trimester of pregnancy). Participants will complete an Epworth sleepiness scale questionnaire and the STOP questions before having their BMI, age and neck circumference documented. A STOPBANG score and Modified STOPBANG score (substitute tired question with Epworth >10) will be calculated. All participants will then take a Rad8 pulse oximeter home to record their overnight pulse rate and oxygen saturations. The oximetry results will be analysed by a respiratory physiologist and the oxygen desaturation index will be calculated. A statistician will analyse the results to determine if there is a relationship between STOPBANG score or Modified STOPBANG score and likelihood of the pregnant women having OSA. In a secondary analysis we will then see if any individual elements of STOPBANG can be used to predict OSA.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Body mass index ≥ 40 at first midwife appointment
* Women ≥ 18 years of age

Exclusion Criteria:

* Pre-existing obstructive sleep apnoea on treatment
* Pre-existing restrictive or obstructive respiratory disease
* Women with another cause of sleep apnoea (e.g. central sleep apnoea)
* Women under 18 years of age
* Women who do not provide or refuse consent
* Women lacking capacity to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women booked to deliver at Sunderland Royal Hospital who have a body mass index ≥40 at their first midwife appointment.
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Obstructive Sleep Apnoea | Between weeks 17-28 of pregnancy
  Oxygen desaturation index (4% from baseline) > 5 per hour

SECONDARY OUTCOMES:
STOPBANG score | Between weeks 17-28 of pregnancy
  Snore, Tired, Observed to Stop Breathing, high blood Pressure, BMI, Age, Neck circumference, Gender
Modified STOPBANG score | Between weeks 17-28 of pregnancy
  Snore, Epworth > 10, Observed to Stop Breathing, high blood Pressure, BMI, Age, Neck circumference, Gender

CONTACTS AND LOCATIONS:
Overall Officials: Sean Cope, MBBS, Principal Investigator — Consultant Anaesthetist
Locations (1):
- Sunderland Royal Hospital, Sunderland, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pearson F, Batterham AM, Cope S. The STOP-Bang Questionnaire as a Screening Tool for Obstructive Sleep Apnea in Pregnancy. J Clin Sleep Med. 2019 May 15;15(5):705-710. doi: 10.5664/jcsm.7754. PMID 31053210
- See also: Information about STOPBANG validation — http://www.stopbang.ca/publication/validation.php